CLINICAL TRIAL: NCT00302874
Title: In-Hospital Hyperglycemia: Effects of Treatment on Glycemic Control and Clinical Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: gil362-HMO-CTIL
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2002-10

CONDITIONS: Diabetes; Hyperglycemia
Keywords: diabetes; hyperglycemia; hospital; medicine ward
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

INTERVENTIONS:
Behavioral: Implementation of a protocol for treatment of hyperglycemia

SUMMARY:
To improve glycemic control of inpatients admitted to the internal medicine wards, the researchers generated a protocol based on intensive insulin treatment for use in all inpatients with hyperglycemia.

The researchers hypothesize that intensive insulin treatment will improve the glycemic control and the outcome of hospitalized patients.

Study Information:

* All patients with a history of diabetes admitted to the internal medicine ward were enrolled in the study.
* At baseline, demographic and clinical information were obtained, including information necessary to determine the severity of the illness. Venous capillary blood glucose levels were checked 4 times a day by glucometer.
* During the pre-intervention period, patients were treated according to the common practice in the hospital without any intervention. The study team collected the baseline data on the glycemic control and treatment of patients admitted with hyperglycemia.
* During the intervention period, the study team visited the ward daily and guided the medical staff as to the use of the treatment protocol.
* During the post-intervention period, the study team collected the data without active intervention in the implementation of the protocol.
* Data was collected on the mode of treatment and glycemic control of all hyperglycemic patients throughout the study. The incidence of hypoglycemia, complications (myocardial infarction, stroke, infections), mortality, transfer to intensive care unit (ICU), length of hospitalization, and disposition at discharge were noted.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the internal medicine ward with hyperglycemia

Exclusion Criteria:

* Patients admitted due to hypoglycemia, hyperosmolar state, and ketoacidosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2003-02; Study Completion 2004-10

PRIMARY OUTCOMES:
Mean blood glucose during hospitalization

SECONDARY OUTCOMES:
Hypoglycemic events
Length of in-hospital stay
Infections
Complications (myocardial infarction, stroke)
Disposition at discharge (home, nursing home)

CONTACTS AND LOCATIONS:
Overall Officials: Gil Leibowitz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel